CLINICAL TRIAL: NCT02787954
Title: Prospective Evaluation of Tumor Response to Cancer Treatment Therapies
Brief Title: Prospective Tumor Response Evaluation
Acronym: Liver
Status: Terminated | Type: Observational
Why Stopped: PI transferred to another institution and did not take this study with him.
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Sponsor
Other Study IDs: HSC-MS-14-0761
Record Dates: First submitted 2016-05-26; First posted 2016-06-01 (Estimated); Last update posted 2018-10-18 (Actual); Status verified 2018-10

CONDITIONS: Hepatocellular Cancer; Metastatic Liver Cancer
MeSH Terms: conditions — Liver Neoplasms | interventions — Yttrium-90; Electroporation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Biopsy liver tumor samples and blood tumor samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Transcatheter Chemoembolization or TACE: A technique called transcatheter chemoembolization (TACE) is used for some patients with liver cancer that cannot be treated surgically. The procedure is a way of delivering cancer treatment directly to a tumor through minimally-invasive means.
  Interventions: Procedure: TACE
- Yittrium 90 or Y-90: Radioembolization is a minimally invasive procedure that combines embolization and radiation therapy to treat liver cancer. Tiny glass or resin beads filled with the radioactive isotope yttrium Y-90 are placed inside the blood vessels that feed a tumor. This blocks the supply of blood to the cancer cells and delivers a high dose of radiation to the tumor while sparing normal tissue.
  Interventions: Procedure: Y-90
- Microwave Ablation or MWA: Microwave ablation (MWA), destroys liver tumors using heat generated by microwave energy. A CT scan or ultrasonic guidance is used to pinpoint the exact location of the tumor. A thin antenna, which emits microwaves, is then inserted into the tumor. The probe produces intense heat that ablates (destroys) tumor tissue, often within 10 minutes.
  Interventions: Procedure: MWA
- electroporation: Irreversible electroporation (IRE) is a nonthermal method of destroying the cell. A cell is subjected to a powerful electrical field using high-voltage direct current (up to 3 kV); this creates multiple holes in the cell membrane and irreversibly damages the cell's homeostasis mechanism, leading to instant cell death.
  Interventions: Procedure: IRE

INTERVENTIONS:
Procedure: TACE — Procedure for giving chemotherapy directly to tumor cells.
  Other Names: Transcatheter arterial chemoembolization
  Groups: Transcatheter Chemoembolization or TACE
Procedure: Y-90 — Using a combination of radiation and chemotherapy directly on the tumor cells to cause cell death.
  Other Names: Yittrium 90
  Groups: Yittrium 90 or Y-90
Procedure: MWA — Using heat to kill tumor cells.
  Other Names: Microwave Ablation
  Groups: Microwave Ablation or MWA
Procedure: IRE — Using energy to disrupt tumor cell activity, thereby causing cellular death.
  Other Names: Irreversible Electroporation
  Groups: electroporation

SUMMARY:
The purpose of this study is to determine if MRI imaging can detect genetic, proteomic, and metabolomic characteristics of liver tumors. The study also aims to determine if these imaging characteristics are correlated with clinical outcomes.

DETAILED DESCRIPTION:
For each treatment arm, pre-procedural MRI and post procedural MRI will be obtained. Pre-procedural biopsies will be obtained, if possible. Pretreatment genetic expression, proteomic, or metabolomic patterns from the tumor samples will be assessed. Imaging characteristics from tumors will be extracted using automated software-the study will apply a computational analysis system with the capability to extract and analyze imaging characteristics and correlate them to genetic expression, proteomic, and metabolomic tumor characteristics. Imaging findings will be correlated to clinical outcomes and genetic, proteomic, and metabolomic findings to determine association. Imaging findings and genomic, proteomic, and metabolomic tumor characteristics will be correlated to clinical outcomes (time to recurrence, overall survival, 3-month, 6-month, and 1-year survival).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis or suspicion of primary or metastatic liver cancer deemed eligible for TACE, Y-90, percutaneous ablation, and /or electroporation.

Exclusion Criteria:

* Any reason MRI cannot be obtained.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with primary or metastatic liver cancer, who are deemed candidates for TACE, electroporation, MWA, or Y90 will be enrolled. The patients will be recruited from medical oncology, surgical oncology, gastroenterology, and transplant surgery services.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Time to progression | 1 month to 3 years
  Time from initial treatment to progression as defined by RECIST criteria.

SECONDARY OUTCOMES:
1 year survival | 1 year
  Number of patients alive 1 year after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Derek L West, MD, Principal Investigator — University of Texas Healtlh Science Center at Houston
Locations (1):
- University of Texas Health Science Center Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Forner A, Llovet JM, Bruix J. Hepatocellular carcinoma. Lancet. 2012 Mar 31;379(9822):1245-55. doi: 10.1016/S0140-6736(11)61347-0. Epub 2012 Feb 20. PMID 22353262
- [Background] Gu L, Liu H, Fan L, Lv Y, Cui Z, Luo Y, Liu Y, Li G, Li C, Ma J. Treatment outcomes of transcatheter arterial chemoembolization combined with local ablative therapy versus monotherapy in hepatocellular carcinoma: a meta-analysis. J Cancer Res Clin Oncol. 2014 Feb;140(2):199-210. doi: 10.1007/s00432-013-1528-8. PMID 24077865
- [Background] Raoul JL, Gilabert M, Piana G. How to define transarterial chemoembolization failure or refractoriness: a European perspective. Liver Cancer. 2014 May;3(2):119-24. doi: 10.1159/000343867. PMID 24945002
- [Background] Assumpcao L, Choti M, Pawlik TM, Gecshwind JF, Kamel IR. Functional MR imaging as a new paradigm for image guidance. Abdom Imaging. 2009 Nov;34(6):675-85. doi: 10.1007/s00261-008-9481-8. Epub 2008 Dec 2. PMID 19048335
- [Background] Bian DJ, Xiao EH, Hu DX, Chen XY, Situ WJ, Yuan SW, Sun JL, Yang LP. Magnetic resonance spectroscopy on hepatocellular carcinoma after transcatheter arterial chemoembolization. Chin J Cancer. 2010 Feb;29(2):198-201. PMID 20109351
- [Background] Minami Y, Kudo M. Therapeutic response assessment of transcatheter arterial chemoembolization for hepatocellular carcinoma: ultrasonography, CT and MR imaging. Oncology. 2013;84 Suppl 1:58-63. doi: 10.1159/000345891. Epub 2013 Feb 20. PMID 23428860
- [Background] Karlo CA, Di Paolo PL, Chaim J, Hakimi AA, Ostrovnaya I, Russo P, Hricak H, Motzer R, Hsieh JJ, Akin O. Radiogenomics of clear cell renal cell carcinoma: associations between CT imaging features and mutations. Radiology. 2014 Feb;270(2):464-71. doi: 10.1148/radiol.13130663. Epub 2013 Oct 28. PMID 24029645